CLINICAL TRIAL: NCT04981171
Title: Efficacy and Safety of Electro-thumbtack Needle Therapy for Patients With Chronic Neck Pain: a Randomized, Placebo-controlled Trial
Brief Title: Electro-thumbtack Needle Therapy for Chronic Neck Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shi Hangyu (Other)
Responsible Party: Sponsor-Investigator, Shi Hangyu, Principal Investigator, Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Organization: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2021-039-KY-01
Record Dates: First submitted 2021-07-18; First posted 2021-07-28 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Neck Pain
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Electro-thumbtack Needle Therapy (ETN) group (Experimental): Electro-thumbtack needles (0.25×2 mm) will be inserted into acupoints of Dazhui (GV14), bilateral Wangu (GB12), bilateral cervical Jiaji (at C4 and C6 level), two Ashi points and bilateral Houxi (SI3) after sterilization. Then apply the gel electrodes and stimulation devices, turn on the device to produce a proper electric stimulation that the participant can tolerate.
  Interventions: Procedure: Electro-thumbtack Needle Therapy
- Sham Electro-thumbtack Needle Therapy (ETN) group (Sham Comparator): Sham electro-thumbtack needles (0.25×0.2 mm) which are specially produced have blunt tips instead of sharp needle tip. They will be taped on acupoints of Dazhui (GV14), bilateral Wangu (GB12), bilateral cervical Jiaji (at C4 and C6 level), two Ashi points and bilateral Houxi (SI3) after sterilization. Then apply the gel electrodes and stimulation devices, produce a minimal level of electric stimulation for 30 seconds before turning off the device.
  Interventions: Procedure: Sham electro-thumbtack needle therapy

INTERVENTIONS:
Procedure: Electro-thumbtack Needle Therapy — Each treatment session starts with sterilizing acupoints. Dazhui (GV14), bilateral Wangu (GB12), bilateral cervical Jiaji (at C4 and C6 level), two Ashi points and bilateral Houxi (SI3) have been selected in accordance with the principle of acupuncture prescription making and the consensus of experts on treating neck pain. Electro-thumbtack needles (0.25×2 mm) will be held by the acupuncturist between thumb and forefinger, vertically inserted into skin instantly and taped well on skin. Then assemble the gel electrodes to the surface of the conductive adhesive tape, also assemble the portable stimulation devices, adjust the current intensity from level 1 to a proper level that the participant can tolerate. Participants will receive three 30-min treatment sessions per week every other day for 4 consecutive weeks.
  Other Names: ETN
  Arms: Electro-thumbtack Needle Therapy (ETN) group
Procedure: Sham electro-thumbtack needle therapy — Each treatment session starts with sterilizing acupoints. Sham electro-thumbtack needles (0.25×0.2 mm) will be held by the acupuncturist between thumb and forefinger, taped well on skin without penetration. The adhesive tape of needles are also produced with conductive material, after assembling the gel electrodes and the portable stimulation devices, adjust the current intensity to level 1 for a minimal stimulus which will last for only 30 seconds. By this time the acupuncturist will turn the device off to cut the current. Participants will receive three 30-min treatment sessions per week every other day for 4 consecutive weeks.
  Other Names: Sham ETN
  Arms: Sham Electro-thumbtack Needle Therapy (ETN) group

SUMMARY:
This prospective trial will be a single-center, participant-blinded, randomized controlled trial. It is reported in previous studies that both acupuncture and transcutaneous electrical nerve stimulation are effective in reducing neck pain comparing to placebo or exercise. Taking into account the convenience of electro-thumbtack needle therapy shown in clinical practice, this study aims to evaluate the efficacy and safety of electro-thumbtack needle therapy for alleviating chronic neck pain compared with sham electro-thumbtack needle therapy.

DETAILED DESCRIPTION:
Chronic neck pain is a commonly experienced symptom that often influences work efficiency and life satisfaction for years. A total of 180 participants suffering mechanical chronic neck pain will be recruited and randomized into either electro-thumbtack needle therapy group or sham electro-thumbtack needle therapy group. All participants will receive the standardized neck exercise instruction at their first treatment session and will be asked to perform the exercise once every day during 4-week treatment. All assessments will be performed by the assessor and the assessment results will be all kept from the acupuncturist. The statistician will be involved in neither assessment nor treatment and will be blinded regarding intervention group code.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with neck pain with headaches or neck pain with movement coordination impairments according to the Orthopaedic Section of the American Physical Therapy Association (APTA);
2. Aaged 18-65 years;
3. History of neck pain for at least 3 months;
4. A score of ≥4 in Numerical Rating Scale for neck pain (NRS-NP) assessing the average neck pain intensity over last 7 days until the day of recruitment.

Exclusion Criteria:

1. Diagnosed with neck pain with mobility deficits or neck pain with radiating pain according to the Orthopaedic Section, APTA;
2. Known specific reason leading to neck pain such as tumor, immune disease, endocrine and metabolic disorders, neurological abnormalities, cervical vertebra fracture, cervical dislocation;
3. Acute neck pain or neck pain with radiating pain or upper limb symptoms;
4. Neck pain with sensory or motor disturbance;
5. Prior cervical spine surgery or congenital abnormalities;
6. Experiencing medical dispute litigation;
7. Have received acupuncture in last 30 days;
8. In need of analgesic, muscle relaxant, hormones, or bearing greater pain from another area;
9. Allergic to metal or adhesive tape, or carrying cardiac pacemaker, or skin damaged at selected acupoints;
10. Disable to communicate or critically ill;
11. Drug or alcohol dependent;
12. Currently or planning to be pregnant.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2022-04-03 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with an at least 50% decrease in NRS-NP from baseline. | week 4
  Rate pain intensity by 11 numbers from 0 (no pain at all) to 10 (worst pain imaginable)

SECONDARY OUTCOMES:
Change of NRS-NP from baseline. | week 4, 16, 28
  Rate pain intensity by 11 numbers from 0 (no pain at all) to 10 (worst pain imaginable)
Proportion of participants with an at least 50% decrease in NRS-NP from baseline. | week 16, 28
  Rate pain intensity by 11 numbers from 0 (no pain at all) to 10 (worst pain imaginable)
Proportion of participants with an at least 30% decrease in NRS-NP from baseline. | week 4, 16, 28
  Rate pain intensity by 11 numbers from 0 (no pain at all) to 10 (worst pain imaginable)
Change of NPQ from baseline. | week 4, 16, 28
  NPQ is a validated questionnaire to learn about the quality and the duration of neck pain and the difficulty coping with chores because of the pain. It contains 9 questions, each ranging from 0 to 4. The total score will be converted to NPQ percentage score (divided by 36 for people who drive and by 32 for those who don't), which ranges from 0 to 100%. High scores indicate worse condition.
Proportion of participants with an at least 25% decrease in NPQ from baseline and a "better" or "much better" for global effectiveness rating. | week 4, 16, 28
  NPQ is a validated questionnaire to learn about the quality and the duration of neck pain and the difficulty coping with chores because of the pain. It contains 9 questions, each ranging from 0 to 4. The total score will be converted to NPQ percentage score (divided by 36 for people who drive and by 32 for those who don't), which ranges from 0 to 100%. High scores indicate worse condition.
Change of NDI from baseline. | week 4, 16, 28
  NDI is a widely used instrument to measure self-reporting disability due to neck pain. It consists of 10 items scored with an ordinal scale from 0-5. The total score ranges from 0-50. Higher scores indicate greater functional limitation. The translated simplified-Chinese version of NDI has been shown to be a responsive and valid measurement for simplified-Chinese speaking patients.
Proportion of participants with an at least 10-point decrease in NDI from baseline. | week 4, 16, 28
  NDI is a widely used instrument to measure self-reporting disability due to neck pain. It consists of 10 items scored with an ordinal scale from 0-5. The total score ranges from 0-50. Higher scores indicate greater functional limitation. The translated simplified-Chinese version of NDI has been shown to be a responsive and valid measurement for simplified-Chinese speaking patients.
Degree of PGIC. | week 4, 28
  Characterize the participants' overall satisfaction and personal feelings about treatment delivery. The options are ranking from "very much worse" to "very much improved" for patients to define their overall status compared with the start of the study.

OTHER OUTCOMES:
Self-expectation assessment. | baseline
  Participants will be asked "How do you think your neck pain will be after 4 weeks?" for self-expectation, the answers are "worse", "unchanged", "no idea", "better", "much better".
Preference of ETN assessment. | baseline
  Participants will be asked"Do you think ETN will be effective for chronic neck pain?" for preference of ETN, the answers are "not effective", "little effective", "not sure", "effective", "very effective".
Blinding assessment. | week 4
  All participants will be told before allocation that insertion is deeper in ETN group and shallower in sham ETN group, the electric stimulation is weak or just about to feel in both groups. After treatments finished, they will be asked "Do you think you have received ETN in the past weeks?", the answers are "Yes", "No" or "Unclear".
Proportion of participants taking rescue medication. | week 0 to 28
  Any other therapy will be discouraged during this trial. If the neck pain occurs heavily or unbearably, acetaminophen (sustained release type, 500 mg/T) will be provided as rescue medication.
Total days of participants demanding rescue medication. | week 0 to 28
  Any other therapy will be discouraged during this trial. If the neck pain occurs heavily or unbearably, acetaminophen (sustained release type, 500 mg/T) will be provided as rescue medication.

CONTACTS AND LOCATIONS:
Overall Officials: Hangyu Shi, Principal Investigator — Guang'anmen Hospital of China Academy of Chinese Medical Sciences

REFERENCES:
- [Derived] Shi H, Wang X, Yan Y, Zhu L, Chen Y, Gao S, Liu Z. Efficacy and Safety of Electro-Thumbtack Needle Therapy for Patients With Chronic Neck Pain: Protocol for a Randomized, Sham-Controlled Trial. Front Med (Lausanne). 2022 Apr 29;9:872362. doi: 10.3389/fmed.2022.872362. eCollection 2022. PMID 35572961